CLINICAL TRIAL: NCT04180592
Title: Real Time MRI Fused to Cone Beam CT Guided Biopsies of the Prostate: The Safety and Feasibility of a Novel Method of Prostate Biopsy.
Brief Title: Real Time MRI Fused to Cone Beam CT Guided Biopsies of the Prostate.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Jason Izard, Department of Urology, Assistant Professor, Queen's University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 6018147
Record Dates: First submitted 2019-11-20; First posted 2019-11-27 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Prostate Cancer
Keywords: MRI; Prostate Biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized cross-over designed trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT Fusion Biopsy + Transrectal U/S Guided Prostate Biopsy (Experimental): All patients will receive both a CT fusion biopsy and a standard TRUSP biopsy. They will be randomized to which is received first, followed by receipt of the alternative procedure.
  Interventions: Procedure: CT Fusion + Transrectal U/S Guided Prostate Biopsy
- Transrectal U/S Guided Prostate Biopsy + CT Fusion Biopsy (Other): All patients will receive both a CT fusion biopsy and a standard TRUSP biopsy. They will be randomized to which is received first, followed by receipt of the alternative procedure.
  Interventions: Procedure: CT Fusion + Transrectal U/S Guided Prostate Biopsy

INTERVENTIONS:
Procedure: CT Fusion + Transrectal U/S Guided Prostate Biopsy — All patients will receive both a CT fusion biopsy and a standard TRUSP biopsy. They will be randomized to which is received first, followed by receipt of the alternative procedure.

SUMMARY:
The purpose of this study is to investigate a novel method of prostate biopsy using a computerized guidance system to accurately target lesions within the prostate. This method of prostate biopsy involves using a computerized technology that permits a lesion detected on MRI to be projected by a computer into 3 dimensions on a patient's CT scan. A CT guided biopsy can then be performed where a needle is advanced into the patient, where the computer has projected the image of the tumor that cannot normally be seen on CT. This is a randomized, cross over designed trial to compare this new method of prostate biopsy to the currently employed standard transrectal ultrasound guided prostate (TRUSP) biopsy technique.

DETAILED DESCRIPTION:
This will be a prospective randomized controlled trial using a cross over design. Patients will serve as their own controls and undergo both TRUSP biopsy (standard of care) and mpMRI fused to cone beam CT guided biopsy of the prostate. The procedures and recovery will follow the identical standardized care pathway that is currently used for TRUSP biopsies. A total of 20 patients will be recruited

Patients will be randomized to receive either TRUSP biopsy or cone beam CT guided biopsy first, followed by the alternative procedure. Following the initial biopsy procedure the patients will fill out a short pain score. They will then recover in the radiology suite for a period of one hour. Following a one hour recovery period the patient will subsequently undergo the alternative biopsy procedure. They will then fill out a second pain score with two additional questions asking the patient to compare the two biopsy approaches with respect to comfort and preference using a 7 point Likert scale. Specimens will be sent to pathology separately to detect differences in diagnostic yield between the two biopsy approaches. In order to minimize inter-operator variability in outcomes, Dr. Menard will perform all biopsies regardless of approach.

An interim analysis after 10 patients will be performed. The study will be terminated early if:

1. No TRUSP biopsy detects any form of prostate cancer
2. No cone beam CT guided biopsy detects any form of prostate cancer.
3. Average pain scores between biopsy approaches differ by more than 4 points on the Universal Pain Assessment scale.
4. 3 or more patients suffer any of:

   1. Immediate procedure related complications
   2. 30 day return to the emergency room
   3. 30 day hospital admission

Measures

Feasibility:

Patients will be considered to have clinically significant prostate cancer based on their PI-RADS score 4 or 5. The ability of TRUSP biopsy and cone beam CT guided biopsy to detect any form of prostate cancer as well as clinically significant prostate cancer (defined as prostate cancer with a Gleason score ≥7) will serve as the primary outcome measures.

Safety:

Immediate procedure related complications, 30 day return to the ER and 30 day hospital admission rates will be recorded. Immediate procedure related complications will be documented at the time of the procedure. The 30 day return to the ER and hospital admission rates will be documented at the participant's followup appointment. Complication rates will reflect the total combined complication rate. This can be compared against the known Ontario province rates to ensure that the addition of cone beam CT guided biopsy does not provide for additive morbidity.

Tolerability:

Patients will fill out the Universal Pain Assessment Tool after each procedure. After both procedures are completed, patients will fill out two questions utilizing a 7 point Likert scale on preference and comfort between the two biopsy approaches.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be eligible for enrollment if they have both of:

  1. Lesion in the prostate on mpMRI that is highly likely to be clinically significant prostate cancer based on the PI-RADS version 2 score (PI-RADS score of 4 or 5).
  2. A previous negative TRUSP biopsy or previous TRUSP biopsy showing atypical small acinar proliferation, high grade prostatic intraepithelial neoplasia or low volume Gleason 6 disease (low risk disease) all of which are incongruent with the high PI-RADS score of the mpMRI lesion.

Exclusion Criteria:

1. Uncorrected coagulopathy.
2. Active, untreated urinary tract infection.
3. Inability to access the rectum in order to perform TRUSP biopsy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Accuracy of CT fusion biopsy [number of biopsies that show clinically significant prostate cancer] | Day 0
  Patients will be considered to have clinically significant prostate cancer based on their PI-RADS score 4 or 5. The ability of TRUSP biopsy and cone beam CT guided biopsy to detect any form of prostate cancer as well as clinically significant prostate cancer (defined as prostate cancer with a Gleason score ≥7) will serve as the primary outcome measures.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]). | 0 Day and at 30 day
  Immediate procedure related complications will be documented at the time of procedures. The 30 day return to the ER and hospital admission rates will be documented at the participant's following appointment.
Tolerability of CT fusion biopsy | Day 0
  Patients will fill out the 0-10 point Universal Pain Assessment Tool after each procedure where 0 is no pain and 10 is the worst pain possible. After both procedures are completed, patients will also fill out two questions utilizing a 1-7 point Likert scale on preference and comfort between the two biopsy approaches where 1 represents rectum biopsy and 7 represents buttock muscle biopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada